CLINICAL TRIAL: NCT01215903
Title: The Beneficial Effects of Fish Nutrients on the Obesity-linked Metabolic Syndrome and Cardiovascular Risk Profile
Brief Title: Fish Gelatin Supplement and Omega-3 Supplement in Obese or Overweight Subjects With Insulin Resistance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Advance Foods and Materials Network (Other); Institut des Nutraceutiques et Aliments fonctionnels, Quebec (Clinical nutrition facilities) (Unknown); University of Guelph (Other); Ocean Nutrition Canada, Halifax (in-kind support: omega-3 supplements) (Unknown); Kenney & Ross (Other)
Responsible Party: Helene Jacques, PhD, Laval University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: SIRUL-85742
Record Dates: First submitted 2010-10-05; First posted 2010-10-07 (Estimated); Last update posted 2010-10-25 (Estimated); Status verified 2010-10

CONDITIONS: Insulin Resistance; Type 2 Diabetes
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2 | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fish gelatin and omega-3 (Experimental)
  Interventions: Dietary Supplement: Fish gelatin and omega-3 polyunsaturated fatty acid
- Omega-3 (Experimental)
  Interventions: Dietary Supplement: Omega-3 polyunsaturated fatty acid

INTERVENTIONS:
Dietary Supplement: Fish gelatin and omega-3 polyunsaturated fatty acid
  Arms: Fish gelatin and omega-3
Dietary Supplement: Omega-3 polyunsaturated fatty acid
  Arms: Omega-3

SUMMARY:
The present study was conducted to test whether a fish gelatin supplement combined with an omega-3 polyunsaturated fatty acid supplement can exert beneficial and sex-specific effects on insulin sensitivity, glucose tolerance, indicators of insulin secretion, blood pressure, lipid metabolism, inflammation and energy intake in obese or overweight insulin-resistant men and women. The investigators hypothesis is that fish gelatin improves insulin sensitivity, glucose tolerance, lipid profile and reduces inflammation in obese or overweight insulin-resistant men and women.

DETAILED DESCRIPTION:
An important number of recent epidemiological studies have demonstrated the beneficial effects of marine omega-3 polyunsaturated fatty acids (n-3 PUFA) on cardiovascular disease risk factors such as reduced triglycerides, decreased platelet aggregation, plaque stabilization, antiarrhythmic effects, and reduced blood pressure. Dietary fish protein has also been shown to improve insulin sensitivity by 30% in insulin-resistant obese or overweight human subjects. In addition, an increasing number of studies describe and demonstrate the physiological and metabolic variations between men and women in regard to CVD and their risk factors, including type 2 diabetes, but the data are still limited. In agreement with the recent findings, this study was conducted to evaluate the combined and synergistic effects of omega-3 and fish protein supplements on insulin sensitivity, blood pressure, lipid metabolism and inflammation in obese or overweight insulin-resistant men and women having some or all the metabolic syndrome criteria including a deteriorated lipid profile, high blood pressure and high waist circumference in a free living situation.

ELIGIBILITY:
Inclusion Criteria:

* overweight or obese (body mass index [BMI] between 25 and 40kg/m2)
* fasting plasma glucose below 7.0mmol/L and 2-h plasma glucose below 11.1mmol/L
* fasting plasma insulin above 90pmol/L

Exclusion Criteria:

* Diabetes, chronic, metabolic or acute disease
* Major surgery within the last 3 months
* Significant weight loss (±10%) within the last 6 months
* Any medication-taking known to affect lipid of glucose metabolism
* Allergy, intolerance or dislike of fish
* Smokers

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-11; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | At 8 weeks
Plasma lipids and lipoproteins | at 8 weeks
Blood pressure | At 8 weeks
Plasma and serum inflammatory markers | At 8 weeks

SECONDARY OUTCOMES:
Glucose tolerance | At 8 weeks
Energy intake | At 8 weeks
Fatty acids of phospholipids in skeletal muscle | At 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Helene Jacques, PhD, Principal Investigator — Laval University; Andre Marette, PhD, Principal Investigator — Laval University; John S Weisnagel, MD/FRCPC, Principal Investigator — Laval University
Locations (1):
- Laval University, Québec, Quebec, Canada